CLINICAL TRIAL: NCT04386772
Title: Preoperative Portal Vein Embolization Using Coils Plus TAGM vs Multiple Coils for Patients With Perihilar Cholangiocarcinoma or Hepatocellular Carcinoma: a Randomized Controlled Study
Brief Title: Portal Vein Embolization Using Coils Plus TAGM vs Multiple Coils for Patients With Perihilar Cholangiocarcinoma or Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor and Chief Surgeon, Principal Investigator, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2018-02-024
Record Dates: First submitted 2020-05-01; First posted 2020-05-13 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Portal Vein Occlusion; Cholangiocarcinoma, Perihilar; Hepatocellular Carcinoma; Liver; Hypertrophy, Acute
Keywords: Portal vein embolization; Trisacryl gelatin microspheres; Coils; Major hepatectomy; Liver hypertrophy
MeSH Terms: conditions — Klatskin Tumor; Carcinoma, Hepatocellular; Hypertrophy | interventions — trisacryl gelatin microspheres

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVE with coils plus TAGM (Experimental): PVE with coils proximally plus TAGM distally and subsequent major hepatectomy
  Interventions: Procedure: PVE with coils plus TAGM
- PVE with multiple coils (Active Comparator): PVE with multiple coils and subsequent major hepatectomy
  Interventions: Procedure: PVE with multiple coils

INTERVENTIONS:
Procedure: PVE with coils plus TAGM — PVE with TAGM distally and coils proximally and subsequent scheduled major hepatectomy. Sequential transcatheter arterial chemoembolization and PVE for patients with HCC. Selective biliary drainage on future liver remnant (FLR) side for patients with pCCA when obstructive jaundice is present.
  Arms: PVE with coils plus TAGM
Procedure: PVE with multiple coils — Procedure: PVE with multiple coils PVE with multiple coils proximally and distally and subsequent scheduled major hepatectomy. Sequential transcatheter arterial chemoembolization and PVE for patients with HCC. Selective biliary drainage on FLR side for patients with pCCA when obstructive jaundice is present.
  Arms: PVE with multiple coils

SUMMARY:
The aim of this study is to investigate the differences of safety and liver hypertrophy between portal vein embolization (PVE) using coils plus tris-acryl gelatin microspheres (TAGM) and multiple coils in patients with perihilar cholangiocarcinoma (pCCA) or with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Perihilar cholangiocarcinoma (pCCA) and hepatocellular carcinoma (HCC) both are common primary hepatobiliary tumors, which often require extensive hepatic resection and challenge perioperative management as surgery remains the only chance of long-term survival for such patients. PVE induces effective hypertrophy on one side of the liver parenchyma ahead of a planned liver resection of the other side which becomes atrophic.

Technically, the percutaneous transhepatic approach becomes the standard of care for PVE. PVEs themselves with different embolization materials could vary in the degree of liver hypertrophy, though some techniques, such as TAE, HVE and stem cell, have been already used in combination with PVE and could promote the hypertrophy. Several aspects on the use of PVE are insufficiently studied and most recommendations are based on low-grade evidence. Large clinical studies that compare the effect of different embolic materials on the hypertrophy response are lacking. PVE using multiple coils to completely occlude all the target segmental and sectional branches is a conventional and fundamental approach in our center, which ensured a reliable hypertrophy response with a low PVE-related morbidity and post-hepatectomy liver failure rate in the past decades. PVE using with tris-acryl gelatin microspheres (TAGM) distally and coils proximally, which needs more interventional experience, has become one of standard approaches in our center. However, the study of high-grade evidence regarding the hypertrophy effect of PVE with TAGM and coils is still lacking.

In this randomized study, the investigators aim to compare PVE using TAGM plus coils to PVE using coils alone, in term of PVE-related complications, hypertrophy degree, hepatectomy completion rate, post-hepatectomy liver failure rate, features of immunohistochemical examination on parenchyma, for patients stratified by either pCCA or HCC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and ≤ 70 years of age.
* Diagnosis of pCCA or HCC (through imaging, serology, and/or histological biopsy)
* Performance status: Karnofsky score ≥ 70
* Candidates for right portal vein embolization for potential major hepatectomy with curative intent. Volumetric indication for PVE is less than 40% of standardized FLR.
* Selective biliary drainage on FLR side for patients with pCCA should be performed when total bilirubin level is above 85.5μmol/L or bile duct dilation of FLR presents. Transcatheter arterial chemoembolization should be performed between 1 and 4 weeks before PVE for patients with HCC.
* Criteria of liver function: Child-Pugh A-B7 level, serum total bilirubin < 85.5μmol/L after biliary drainage in pCCA, alanine aminotransferase and aspartate aminotransferase ≤ 3 times the upper limit of normal value.
* Patients who can understand this trial and have signed the informed consent.

Exclusion Criteria:

* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction, which may affect the treatment.
* Patients with a history of any other malignant tumor, or allergic to iodine or gelatin.
* Subjects participating in other clinical trials.
* Platelet count < 80×109/L and/or moderate or severe esophageal varices.
* ICGR15 ≥ 15% for HCC patients
* Obstructive jaundice lasts for >2 months before PVE for pCCA patients.
* Tumor becomes unresectable by local progression and/or distant metastasis presents before PVE.
* Right portal vein is occluded by tumor invasion or embolus before PVE.
* Free portal vein pressure >20 mmHg or porto-hepatic vein fistula at the beginning of PVE procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
PVE related morbidity | During and 2 weeks after PVE procedure
  The rate of major and minor PVE-related complications
Hypertrophy degree of standardized FLR | 2 weeks after PVE procedure
  The difference of standardized FLR ratios before and 2 weeks after PVE

SECONDARY OUTCOMES:
Hepatectomy completion rate | The end of hepatectomy procedure
  The rate of completed major hepatectomy in each Arm group
Liver failure rate after major hepatectomy | 3 months after hepatectomy
  The rate of liver failure measured by 50-50, TB peak 7mg, and ISGLS criteria
Immunohistochemical stainings of liver parenchyma | During (sampling) and immediately after hepatectomy (IHC examination)
  Immunohistochemical stainings of hypertrophic and atrophic parenchyma including anti-albumin, anti-PCNA, TUNEL staining, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Easter hepatobiliary surgery hospital, Shanghai, Shanghai Municipality, China